CLINICAL TRIAL: NCT06706622
Title: Interventional, Randomized, Double-blind, Placebo-controlled, Optional Open-label Extension Trial of Lu AF82422 in Participants With Multiple System Atrophy
Brief Title: A Trial of Amlenetug (Lu AF82422) in Participants With Multiple System Atrophy (MSA)
Acronym: MASCOT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20432A; 2024-517169-18-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple System Atrophy
Keywords: Lu AF82422; MSA; Neurodegenerative Disorder
MeSH Terms: conditions — Multiple System Atrophy; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Amlenetug Low Dose (Experimental): Participants will receive amlenetug by intravenous infusion
  Interventions: Drug: Amlenetug
- Amlenetug High Dose (Experimental): Participants will receive amlenetug by intravenous infusion
  Interventions: Drug: Amlenetug
- Placebo (Placebo Comparator): Participants will receive commercially available saline solution for infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amlenetug — Solution for infusion
  Other Names: Lu AF82422
  Arms: Amlenetug High Dose; Amlenetug Low Dose
Drug: Placebo — Commercially available saline solution
  Arms: Placebo

SUMMARY:
The main goal of this trial is to evaluate the efficacy and safety of amlenetug for the treatment of participants with Multiple System Atrophy (MSA).

DETAILED DESCRIPTION:
This study will consist of a screening period of 10 days up to 6 weeks, a 72-week placebo-controlled period (PCP), and will include a 72-week optional dose-blinded open-label treatment extension (OLE) period. Participants in the PCP will be randomized to amlenetug high dose, amlenetug low dose or placebo (1:1:1). All participants entering the OLE will receive amlenetug during the OLE. Participants will receive intravenous infusions approximately every 4 weeks during both the PCP and OLE.

ELIGIBILITY:
Key Inclusion Criteria:

* The participant has a diagnosis of clinically established multiple system atrophy parkinsonian type (MSA-P) or multiple system atrophy cerebellar type (MSA-C), or clinically probable MSA-P or MSA-C, according to the 2022 Movement Disorders Society (MDS) criteria for the diagnosis of MSA at the Screening Visit.
* The participant had onset of motor MSA symptoms (that is, parkinsonian and/or cerebellar) within 5 years prior to the Screening Visit in the judgement of the investigator.
* The participant has an anticipated survival of >3 years, in the opinion of the investigator, at the Screening Visit.
* The participant has suitable peripheral venous access for investigational medicinal product (IMP) administration and blood sampling.
* The participant has an UMSARS Part I score ≤16 (omitting item 11 on sexual function) at the Screening Visit.

Exclusion Criteria:

* The participant has previously been dosed with amlenetug.
* The participant has taken any active IMP within 3 months or 5 half lives of that product, whichever is longer, prior to the first dose of IMP.
* The participant has 2 or more first degree relatives with a history of MSA.
* The participant, if of MSA-P subtype, has unexplained anosmia (not explained by other common causes such as allergic rhinitis or smoking, nasal structural lesions, or nasal surgery) on olfactory testing at the Screening Visit.
* The participant has evidence (clinically or on magnetic resonance imaging (MRI)) and/or history of any clinically significant disease or condition other than MSA, that is, in the investigator's opinion, likely to affect CNS functioning, e.g., serious neurological disorder, other intracranial or systemic disease.
* The participant has a current diagnosis of movement disorders that could mimic MSA, e.g., Parkinson's disease, dementia with Lewy bodies, essential tremor, progressive supranuclear palsy, spinocerebellar ataxia, spastic paraparesis, corticobasal degeneration, or vascular, pharmacological, or post-encephalitic parkinsonism, per investigator discretion. Participants who have previously been incorrectly diagnosed with Parkinson's disease will not be excluded.

Other protocol-defined inclusion and exclusion criteria apply.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2028-02-17 (Estimated); Study Completion 2029-10-25 (Estimated)

PRIMARY OUTCOMES:
Rest of the World (RoW; All Countries Except European Union [EU] and Japan [JP]) Regional-specific Outcome Measure: Mortality-adjusted Clinical Progression | Baseline up to Week 72
  Mortality-adjusted clinical progression will be assessed by the composite endpoint modified Unified Multiple System Atrophy Rating Scale (mUMSARS) score and time-to-death (any cause).
EU and JP Regional-specific Outcome Measure: Mortality-adjusted Clinical Progression | Baseline up to Week 72
  Mortality-adjusted clinical progression will be assessed by the composite endpoint Unified Multiple System Atrophy Rating Scale (UMSARS) Total Score (TS) and time-to-death (any cause).

SECONDARY OUTCOMES:
RoW Regional-specific Outcome Measure: Mortality-adjusted Clinical Progression | Baseline up to Week 72
  Mortality-adjusted clinical progression will be assessed by the composite endpoint UMSARS TS and time-to-death (any cause).
EU and JP Regional-specific Outcome Measure: Change from Baseline in UMSARS TS | Baseline, Week 72
RoW Regional-specific Outcome Measure: Change from Baseline in UMSARS TS | Baseline, Week 72
Mortality-adjusted Clinical Progression | Baseline up to Week 72
  Mortality-adjusted clinical progression will be assessed by the composite endpoint UMSARS Part I and time-to-death (any cause).
Mortality-adjusted Clinical Progression | Baseline up to Week 72
  Mortality-adjusted clinical progression will be assessed by the composite endpoint UMSARS Part II and time-to-death (any cause).
Change from Baseline in mUMSARS Score | Baseline, Week 72
Change from Baseline in UMSARS Part I Score | Baseline, Week 72
Change from Baseline in UMSARS Part II Score | Baseline, Week 72
Change from Baseline in Clinical Global Impression - Severity of Illness (CGI-S) Score | Baseline, Week 72
Change from Baseline in Patient Global Impression - Severity of Illness (PGI-S) Score | Baseline, Week 72
Change from Baseline in Observer-reported Global Impression-Severity of Illness (OGI-S) Score | Baseline, Week 72
Change from Baseline in UMSARS Part IV Score | Baseline, Week 72
Change from Baseline in Schwab and England Activities of Daily Living (SE-ADL) Score | Baseline, Week 72
Change from Baseline in UMSARS Part I Item 1: Speech Score | Baseline, Week 72
Time to Disability | Baseline up to Week 72
Change from Baseline in EuroQol 5-dimensions, 5-levels (EQ-5D-5L) Domain Score | Baseline, Week 72
Change from Baseline in EQ-5D-5L Visual Analog Scale (VAS) Score | Baseline, Week 72
Change from Baseline in Multiple System Atrophy Quality of Life (MSA-QoL) Questionnaire Domain Scores | Baseline, Week 72
Combined Clinical Progression and Survival Score | Baseline, Week 72
Time from Baseline to Death (Any Cause) | Baseline up to Week 72
Number of Participants with an Absolute Increase in mUMSARS Score of <5, <7, and <9 points | Baseline to Week 72
Number of Participants with an Absolute Increase in UMSARS TS of <16, <21, and <26 Points | Baseline to Week 72
Percentage Change from Baseline in Brain Volume in Brain Regions of Interest (ROIs) | Baseline, Week 72
Area Under the Curve (AUC) of amlenetug | Baseline up to Week 72
Maximum Observed Concentration (Cmax) of Amlenetug | Baseline up to Week 72
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 up to Week 144
Number of Participants with Anti-amlenetug Antibodies (ADAs) | Baseline up to Week 144

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — H. Lundbeck A/S
Locations (74):
- United States (23):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, San Francisco Neurosciences Clinical Research Unit, San Francisco, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Yale New Haven Health, North Haven, Connecticut
  - Parkinson's Disease And Movement Disorder Center Of Boca Raton, Boca Raton, Florida
  - University of Florida Norman Fixel Institute for Neurological Diseases, Gainesville, Florida
  - Indiana Health University, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - QUEST Research Institute, Farmington Hills, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University Nebraska Medical Center, Omaha, Nebraska
  - NYU Medical Center - Dysautonomia center, New York, New York
  - Columbia University Medical Center - The Neurological Institute of New York, New York, New York
  - Cleveland Clinic - Neurological Institute, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center-Cognitive and Movement Disorders Group, Nashville, Tennessee
  - University of Texas Southwestern Medical Center ¿ Multiple System Atrophy Clinic, Dallas, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Inland Northwest Research, Spokane, Washington
- Australia (4):
  - Liverpool Hospital - South Western Sydney Local Health District, Liverpool, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Gold Coast Hospital, Southport, Queensland
  - The Alfred Hospital, Melbourne, Victoria
- Canada (2):
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Toronto Western Hospital (TWH), Toronto, Ontario
- France (7):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Centre Hospitalier Regional Universitaire de Lille - Hopital Roger Salengro, Lille
  - CHU - Hospital de la Timone, Marseille
  - Centre Hospitalier Regional Universitaire (CHRU) Montpellier - Hopital Saint-Eloi Guy de Chauliac, Montpellier
  - Chu De La Pitie-Salpetriere, Paris
  - Unite d'investigation clinique de Neurologie Rez-de-jardin-Bloc Hopital CHU Pontchaillou, Rennes
  - Centre Hospitalier Universitaire de Toulouse - Hopital Purpan, Toulouse
- Germany (6):
  - Movement Disorders Clinic, Beelitz-Heilstätten
  - Universitaetsklinikum Erlangen, Erlangen
  - Curiositas-ad-sanum Beratungs-und Studien GmbH, Haag in Oberbayern
  - Ludwig-Maximilians-Universitat Munchen Klinikum der Universitat - Grosshadern, München
  - Universitaetsklinikum Muenster, Münster
  - University Hospital Tuebingen, Tübingen
- Italy (6):
  - IRCCS Institute of Neurological Sciences of Bologna- Universita di Bologna, Bologna
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - AOU Universita della Campania Luigi Vanvitelli, Napoli
  - A.O.U. Pisana-Ospedale S. Chiara, Pisa
  - Universita Di Salerno Aou San Giovanni Di Dio E Ruggi D'Aragona, Salerno
- Japan (11):
  - National Hospital Organization Higashinagoya National Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Gifu University Hospital, Gifu, Gifu
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Sendai Nishitaga Hospital, Sendai, Miyagi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Center Hospital, National Center of Neurology and Psychiatry, Kodaira-shi, Tokyo
  - Tottori University Hospital, Yonago-shi, Tottori
  - Saitama Medical University Hospital, Iruma-gun
  - Niigata University Medical And Dental Hospital, Niigata
  - Keio University Hospital, Tokyo
- South Korea (3):
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona - Institut Clinic de Neurociencies (ICN), Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona (Spain)
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen del Rocio (HUVR) - Instituto de Biomedicina de Sevilla (IBIS), Seville
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bu..., Valencia
- United Kingdom (6):
  - Salford Royal Hospital, Northern Care Alliance NHS Foundation Trust, Salford, Greater Manchester
  - Nuffield Oxford University and Oxford University Hospital NHS Foundation Trusts-John Radcliffe Ho..., Oxford, Oxfordshire
  - Queen Elizabeth University Hospital - NHS Greater Glasgow & Clyde, Glasgow, Scotland
  - Clinical Ageing Reseach Unit, Newcastle upon Tyne, Tyne and Wear
  - Royal Devon and Exeter Hospital - Royal Devon University Healthcare NHS Foundation Trust, Exeter
  - The National Hospital for Neurology and Neurosurgery, London